CLINICAL TRIAL: NCT03957876
Title: A Phase II Study of CPX-351 as a Novel Therapeutic Approach for Patients With Myelodysplastic Syndromes (MDS) After Hypomethylating Agent Failure
Brief Title: CPX-351 Therapy for MDS After Hypomethylating Agent Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sudipto Mukherjee, Principal Investigator, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2918
Record Dates: First submitted 2019-04-10; First posted 2019-05-21 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — CPX-351; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- intravenous CPX-351 with potential maintenance therapy (Experimental): Single agent CPX-351 administered at the standard FDA approved dose of 44 mg/m2 intravenously on days 1, 3, 5 of the induction cycle. If participants achieve complete remission (CR), complete remission with incomplete count recovery (CRi) or partial remission (PR), they will be eligible to continue on to maintenance therapy, which will consist of CPX351 at a dose of 15.4 mg/m2 every 28 days. Participants can receive up to 4 cycles of maintenance therapy.
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351 — CPX-351 is a liposomal formulation of a fixed combination of the antineoplastic drugs cytarabine and daunorubicin.
  Other Names: (daunorubicin and cytarabine)

SUMMARY:
The purpose of this study is to evaluate the efficacy of treatment with CPX-351 (an FDA approved drug for the treatment of AML) in individuals with MDS while using a new stratification tool to predict outcomes of participants following HMA failure. This approach is intended to gain a better understanding and insight into identifying new opportunities for drug approvals in this setting.

DETAILED DESCRIPTION:
This study will evaluate efficacy of treatment with CPX-351in participants with MDS while using a new stratification tool to predict outcomes of patients following HMA failure in order to gain a better understanding and insight into identifying new opportunities for drug approvals in this setting.

CPX-351is an investigational (experimental) drug for the indication of myelodysplastic syndrome that works by delivering two chemotherapy medications (daunorubicin and cytarabine) together which are then concentrated into the bone marrow (the part of the body that makes blood cells). CPX-351 is experimental because it is not approved by the Food and Drug Administration (FDA) for the indication of myelodysplastic syndrome. This drug is approved by theFDA for the indication of acute myeloid leukemia. One or more of the Investigators conducting this study serve as consultants for the company that makes products used in this study. These financial interests are within permissible limits established by the local institutional Conflict of Interest Policy.

Prior to beginning treatment, all eligible participants will be grouped into low risk versus high risk based on a stratification tool used to determine their disease. Group 1 will be low risk participants and group 2 will be high risk participants. All study participants will get the same study drug, CPX-351. Participants will receive the CPX-351 on days 1, 3 and 5 of the first 28 day cycle. After participants finish the first round of treatment and based on their response they may be eligible for another 4 cycles of treatment. The participant's doctor will inform them if this is an available option when the time comes. Once participant have finished treatment, their doctor will continue observe for side effects and follow their condition for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give voluntary written consent before performance of any study related procedures not part of standard medical care
* Diagnosis of MDS or MDS/MPN according to 2016 WHO criteria12
* Primary therapy failure with either hypomethylating agents (decitabine or azacitidine) defined as:
* Progression (according to 2006 IWG criteria)13 after initiation of azacitidine or decitabine treatment; or
* Failure to achieve complete or partial response or hematological improvement (according to 2006 IWG)13 after at least 4-6 cycles (4-weeks cycle) of azacitidine or decitabine; or
* Relapse after initial complete or partial response or hematological improvement (according to 2006 IWG criteria)13 observed after at least 4 cycles of azacitidine or decitabine.
* Eastern Cooperative Oncology Group (ECOG) Performance Status < 2
* Subjects must have normal organ and marrow function defined as:
* If total bilirubin < 2x upper limit of normal (</= 3 x ULN if considered to be due to leukemic involvement or Gilbert's syndrome) at the discretion of the treating physician following discussion with PI)
* Calculated creatinine clearance value of > 30ml/min AND a serum creatinine < 1.5mg/dL
* LVEF >/= 50%
* Female patients who:
* Are postmenopausal for at least 1 year before the screening visit, OR
* Are surgically sterile, OR
* Agree to practice true abstinence from heterosexual contact or agree to use effective contraception without interruption during the study therapy and 90 days after the last dose
* Male patients who:
* Are surgically sterile, OR
* Agree to practice true abstinence from heterosexual contact or agree to use effective contraception without interruption during the study therapy and 90 days after the last dose

Exclusion Criteria:

* Prior treatment with CPX-351, or known hypersensitivity to CPX-351 or its components.
* Prior treatment with intensive chemotherapy.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that, in the view of the treating physician, would place the participant at an unacceptable risk if he or she were to participate in the study or would prevent that person from giving informed consent.
* Any active malignancy (unrelated, non-hematological malignancy) diagnosed within the past 6 months of starting the study drug (other than curatively treated carcinoma-in-situ of the cervix or non-melanoma skin cancer).
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known history of HIV or active hepatitis B or C.
* Major surgery within 2 weeks prior to study enrollment.
* Pregnant or lactating females
* Male and female patients who are fertile who do not agree to use an effective barrier methods of birth control (i.e. abstinence or 2 forms of contraception) to avoid pregnancy while receiving study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudipto Mukherjee, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The study team does not plan to share IPD collected in this study

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous CPX-351 With Potential Maintenance Therapy
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intravenous CPX-351 With Potential Maintenance Therapy
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of CPX-351 as Measured by Overall Response Rate (ORR)
Description: Efficacy of CPX as measured by ORR as defined by IWG 2006 criteria for MDS participants at end of induction. IWG 2006 responses that must be for at least 4 weeks include Complete Remission (CR), Partial Remission (PR), Marrow CR, Stable Disease (SD), Failure, Relapse after CR or PR (PD), or cytogenetic response. Hematologic Improvement (HI), which must be for at least 8 weeks, includes erythroid response (pretreatment, < 11 g/dL), Platelet response (pretreatment, < 100x109/L), Neutrophil response (pretreatment, < 1 x109/L), or Progression or relapse after HI.
Time Frame: day 28 +/- 7 days of induction
Population: 3 of the 4 participants did not meet evaluable criteria as they did not survive to C1D1 of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous CPX-351 With Potential Maintenance Therapy
Number analyzed (Participants) | 1
Participants
  Complete remission (CR) | 1
  Partial remission (PR) | 0
  Marrow CR | 0
  Stable disease (SD) | 0
  Failure | 0
  Relapse after CR or PR (PD) | 0
  Cytogenetic response | 0

2. Secondary Outcome: Time to Response (TTR) Associated With CPX-351
Description: TTR associated with CPX-351 in participant with MDS at the end of induction. TTR defined by the time between starting the treatment and the time of achieving best response.
Time Frame: day 28 +/- 7 days of induction
Population: 3 additional subjects did not receive study drug (only completed induction phase).
Measure: Number; unit: Days
Arm/Group | Intravenous CPX-351 With Potential Maintenance Therapy
Number analyzed (Participants) | 1
Days | 28

3. Secondary Outcome: Duration of Response (DOR) in Participants Achieving a Response
Description: DOR in participants achieving a response defined by the time between first response (day C1 D28 +/-7 days from induction) and the day of loss of response
Time Frame: up to 1 year after end of treatment
Population: 3 of the 4 participants did not meet evaluable criteria as they did not survive to C1D1 of study.
Measure: Number; unit: days
Arm/Group | Intravenous CPX-351 With Potential Maintenance Therapy
Number analyzed (Participants) | 1
days | 458

4. Secondary Outcome: Event-free Survival (EFS)
Description: EFS probability of all participants enrolled in this trial from start of treatment and up to 1 year after the end of treatment.
Time Frame: up to 1 year after end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous CPX-351 With Potential Maintenance Therapy
Number analyzed (Participants) | 4
Participants | 1

5. Secondary Outcome: Overall Survival (OS)
Description: OS probability of all participants enrolled in this trial from start of treatment and up to 1 year after the end of treatment.
Time Frame: up to 1 year after end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous CPX-351 With Potential Maintenance Therapy
Number analyzed (Participants) | 4
Participants | 1

ADVERSE EVENTS:
Time Frame: 2.5 years or until death, whichever occurs first.
Arm/Group | Intravenous CPX-351 With Potential Maintenance Therapy
All-Cause Mortality (participants affected / at risk) | 4/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous CPX-351 With Potential Maintenance Therapy (N=4)
Anemia (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous CPX-351 With Potential Maintenance Therapy (N=4)
Anemia (Blood and lymphatic system disorders) | 4
Cardiac disorders (Blood and lymphatic system disorders) | 2
Chest pain - cardiac (Blood and lymphatic system disorders) | 1
Febrile neutropenoa (Blood and lymphatic system disorders) | 3
Sinus Tachycardia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Fecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gum bleeding (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 1
Lung infection (Infections and infestations) | 1
Other (Infections and infestations) | 4 — Other, specify (Infection VRE; Infection -- c. difficile; Sputum polymicrobial bacteremia; Bactereia - blood cultures postivie for VRA)
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Sputum pseudomonas (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood biliruib increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decrease (Investigations) | 1
Platelet count decreased (Investigations) | 3
Weight gain (Investigations) | 1
White blood cell descreased (Investigations) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypomagnesmia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Memory Impairment (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination led to a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT03957876/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT03957876/ICF_001.pdf